CLINICAL TRIAL: NCT03760276
Title: A Pilot Study to Evaluate the Appropriateness of the Voriconazole Dosing Regimen Based on the Population Pharmacokinetic Model and the Influence of Sex on the Pharmacokinetics of Voriconazole
Brief Title: A Study to Evaluate the Appropriateness of the Voriconazole Dosing Regimen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, SeungHwan Lee, Clinical Assistant Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Voriconazole_CYP2C19
Record Dates: First submitted 2018-11-23; First posted 2018-11-30 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Fungal Infection
MeSH Terms: conditions — Mycoses | interventions — Voriconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Voriconazole TBD mg tablet orally, every 12 hours for 7 days (Experimental)
  Interventions: Drug: Voriconazole Oral Product (Vfend®)

INTERVENTIONS:
Drug: Voriconazole Oral Product (Vfend®) — To be determined mg of Voriconazole (Vfend®, anti-fungal agent)

SUMMARY:
A pilot study was performed to evaluate the appropriateness of the voriconazole dosing regimen based on the population pharmacokinetic model and the influence of sex on the pharmacokinetics of voriconazole

ELIGIBILITY:
Inclusion Criteria:

* Those who have been informed of the nature of the trial and have voluntarily agreed to participate in this study and have signed an IRB approved consent before all screening tests
* Healthy Korean male and female volunteers aged 20 to 45
* Those with a body weight of 50 kg or more and less than 90 kg and a body mass index (BMI) of 18 or more and less than 27 (BMI(kg/m2) = body weight (kg)/{height(m)}2
* CYP2C19 EM or PM

Exclusion Criteria:

* Subjects with clinical evidence of significant respiratory, circulatory, renal, hepatic, endocrine, blood, neuropsychiatric, skeletal or other chronic diseases, alcohol or drug addiction
* Subjects with a history of gastrointestinal disorders (Crohn's disease, ulcers, acute or chronic pancreatitis, etc.) or gastrointestinal surgery (excluding simple cecal surgery or hernia surgery) that may affect the absorption of the test drug
* Those with a history of substance abuse within the last 2 months
* Those who have taken any prescribed medicines or herbal medicines within 2 weeks prior to the date of the first medicines, or those taking any general medicines (OTC) or vitamin preparations (eligible if the other conditions are reasonable according to the judgment of the investigator)
* Those who donate blood within 30 days before the date of the first dose or who have participated in the clinical study of other clinical trial drugs or marketed drugs within 3 months
* Those who have had significant adverse reactions such as hypersensitivity reactions to azole drugs including drugs for clinical research
* Those who are not planning on or planning to have a pregnancy during the trial and are not able to use a recognized method of contraception (eg, sterilization surgery of the person and partner, intrauterine contraceptive device, or diaphragm contraception (such as diaphragm or condom use)
* Persons who are continuously drinking (21 units / week, 1 unit = 10 g of pure alcohol) or who can not abstain from 3 days before the first dose to the end of the clinical trial
* Those who smoked more than 10 cigarettes per day for the last 3 months or who can not quit smoking 3 days before the first dose
* Those who consume grapefruit / caffeine-containing food within 3 days of the first dose or who cannot be prohibited during the clinical study period
* Screening tests for urine pregnancy (β-hCG) positive or lactating women
* Those with genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
* A person who is found to be unsuitable for participation in clinical research due to safety laboratory results or other reasons

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2018-10-28 (Actual); Study Completion 2018-10-28 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) | Day 1 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours, Day 5 12 hours, Day 6 0, 12 hours, Day 7 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours
  Pharmacokinetic sampling after administration of drugs from day 1 to day 7
Area under the plasma concentration versus time curve from the time of dosing to the last measurable concentration (AUClast) | Day 1 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours, Day 5 12 hours, Day 6 0, 12 hours, Day 7 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours
  Pharmacokinetic sampling after administration of drugs from day 1 to day 7

SECONDARY OUTCOMES:
Genetic polymorphisms of CYP2C9 and CYP3A4 | Day 1 0 hour
  Exploratory evaluation
Hepatic safety marker of miRNA-122 | Day 1 0 hour, Day 5 12 hour, Day 7 12 hour
  Exploratory safety evaluation
Safety and tolerability evaluation by monitoring adverse events (number of subjects and cases) | Day 1 to Day 12
  Safety and tolerability evaluation
Physical examination (list of current medications) | Day 1 to Day 12
  Safety and tolerability evaluation
Physical examination (list of any symptoms or pain) | Day 1 to Day 12
  Safety and tolerability evaluation
Physical examination (Medical and surgical history) | Day 1 to Day 12
  Safety and tolerability evaluation
Evaluation of Vital signs (body temperature °C) | Day 1 to Day 12
  Safety and tolerability evaluation
Evaluation of Vital signs (blood pressure mmHg) | Day 1 to Day 12
  Safety and tolerability evaluation
Evaluation of Vital signs (pulse (heart rate, beats per minute)) | Day 1 to Day 12
  Safety and tolerability evaluation
Evaluation of Vital signs (breathing rate (respiratory rate, beats per minute)) | Day 1 to Day 12
  Safety and tolerability evaluation
Safety and tolerability evaluation by 12-lead ECG (P wave, PR interval, QRS complex, J-point, ST segment, T wave, Corrected QT interval, U wave) | Day 1 to Day 12
  Safety and tolerability evaluation
number of participants with abnormal laboratory values (hematologic, chemical, urine) | Day 1 to Day 12
  Safety and tolerability evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital Clinical Trial Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No